CLINICAL TRIAL: NCT02042508
Title: Evaluation of a Hybrid Prototype Strategy (Electrostimulation of Lower Limb Muscles Associated With Voluntary Strengthening of the Upper Limbs) in Reconditioning to Effort in Patients With Chronic Paraplegia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CASILLAS PARI 2011
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Chronic Paraplegia
MeSH Terms: interventions — Resistance Training

ARMS (1):
- Paraplegic patients (Experimental)
  Interventions: Other: strengthening; Other: hybrid training programme

INTERVENTIONS:
Other: strengthening
Other: hybrid training programme

SUMMARY:
This single-centre study was carried out in collaboration with the Cardiovascular Research Laboratory of Harvard University (Boston, USA). This preliminary study does not include a control group.

The aim of this study was to investigate the effect of a hybrid reconditioning programme (electrostimulation of the lower limb muscles associated with voluntary strengthening of the upper limbs) on a specially developed rowing machine in patients presenting stabilized paraplegia of a traumatic origin. This study will bear on the increase in maximal aerobic capacity (VO2max) between the start and end of the 9-month reconditioning programme.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with paraplegia, ageb between 18 and 45 years
* Body mass index (BMI) between 18.5 and 29.9
* 2 to 15 years after the accident, ASIA A or B, lesion situated between T3 and T12
* Medically stable
* Able to follow instructions
* Persons who have provided written informed consent

Exclusion Criteria:

* Persons without national health insurance cover
* Arterial blood pressure > 140/90 mmHg, arrythmia, heart disease, diabetes, impaired kidney function, cancer
* smoking-induced intoxication,
* Medical treatment for cardiovascular disease or antidepressants
* Orthostatic hypotension with a symptomatic fall in arterial pressure > 30 mmHg in the vertical position
* Grade 2 or more pressure sores
* Other associated neurological diseases (e.g. cerebrovascular accident, peripheral neuropathy, myopathy)
* Any disease affecting the shoulder that may compromise the ability to use the rowing machine.
* Coagulation disorders;
* Presence of an implanted electronic device
* Epilepsy

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-02-02 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max) measured during an incremental maximum effort test | Change from baseline in VO2max at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France